CLINICAL TRIAL: NCT02081482
Title: Study of the Cerebral Metabolism in Patients With Refractory Chronic Cluster Headache Treated by Occipital Nerve Stimulation
Brief Title: Cerebral Metabolism in Patients With Refractory Chronic Cluster Headache Treated by Occipital Nerve Stimulation
Acronym: MET-ONS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-AOI-05
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Refractory Chronic Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- subjects with refractory chronic cluster headache (Experimental): Adult subjects with refractory chronic cluster headache and ONS indication
  Interventions: Radiation: 18F-FDG PET

INTERVENTIONS:
Radiation: 18F-FDG PET

SUMMARY:
The occipital nerve stimulation (ONS) is used to treat patients with refractory primary chronic headache but its mechanism of action (MoA) remains unknown. Different hypothesis have been suggested in particular a specific action on cerebral generators involved in different types of primary headaches or a non specific action on pain modulatory network.

The aim of this study, using the chronic cluster headache as a model, is to determine the changes in cerebral metabolism induced by ONS to precise its MoA in the treatment of primary chronic headache.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* chronic cluster headache (according to the IHS)
* refractory in who a treatment by ONS have been indicated
* patient affiliated at social security,
* informed consent signed

Exclusion Criteria:

* contraindication to MRI
* contraindication to 18F-FDG PET
* women without contraception/pregnant/breast-feeding
* patient non-compliant
* patient on legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of cerebral metabolism | Baseline (before ONS), 1 week after ONS , 3 month after ONS
  Changes of cerebral metabolism associated with ONS efficacy

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU -Hôpital Gabriel Montpied, Clermont-Ferrand
  - Institut des Neurosciences, Marseille
  - Département d'Evaluation et Traitement de la Douleur - Pôle Neurosciences Cliniques - Centre Hospitalo-Universitaire de Nice, Nice
  - Centre d'Urgence Céphalées, Paris